CLINICAL TRIAL: NCT06967051
Title: An Open Label Pilot Study Evaluating the Efficacy of a Smart Phone-based Test on Measuring Pupillary Light Reflex Alterations Following Cannabis Use Healthy in Adults
Brief Title: The Efficacy of a Smart Phone-based Test on Measuring Pupillary Light Reflex Alterations Following Cannabis Use Healthy in Adults
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sobereye Inc. (Industry)
Collaborators: KGK Science Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 24SICFP01
Record Dates: First submitted 2025-04-14; First posted 2025-05-13 (Actual); Last update posted 2025-07-17 (Actual); Status verified 2025-04

CONDITIONS: Cannabis Intoxication; Drug Effects
Keywords: Pupillometer; Cannabis Use; Drug Effects; SOBEREYE; OPTOVERA; Pupillary Light Reflex
MeSH Terms: interventions — Dronabinol

STUDY DESIGN:
Intervention Model Description: Open label pilot study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tetrahydrocannabinol (10 mg) (Experimental): 10 mg of Tetrahydrocannabinol (THC) provided as a softgel capsule.
  Interventions: Drug: Tetrahydrocannabinol (10 mg); Diagnostic Test: Pupillary Light Reflex (PLR) Test; Diagnostic Test: Pupillometer
- Tetrahydrocannabinol (25 mg) (Experimental): 25 mg of THC provided as a softgel capsule.
  Interventions: Drug: Tetrahydrocannabinol (25 mg); Diagnostic Test: Pupillary Light Reflex (PLR) Test; Diagnostic Test: Pupillometer

INTERVENTIONS:
Drug: Tetrahydrocannabinol (10 mg) — 10 mg of Tetrahydrocannabinol (THC) provided as a softgel capsule
  Arms: Tetrahydrocannabinol (10 mg)
Drug: Tetrahydrocannabinol (25 mg) — 25 mg of THC provided as a softgel capsule.
  Arms: Tetrahydrocannabinol (25 mg)
Diagnostic Test: Pupillary Light Reflex (PLR) Test — SOBEREYE OPTOVERA is a portable, non-invasive test that measures the Pupillary Light Reflex (PLR)
Diagnostic Test: Pupillometer — NeuroLight is an automated pupillometer that generates a flash of light and measures the photomotor reflex very accurately.

SUMMARY:
The goal of this open label study is to evaluate the efficacy of smart phone-based test (SOBEREYE OPTOVERA) on measuring pupillary light reflex (PLR) alterations following cannabis use healthy in adults. The main question it aims to answer is:

Can SOBEREYE OPTOVERA detect PLR alterations following cannabis consumption in healthy adults, in comparison to a pupillometer?

Participants will be given two 5 mg capsules to be ingested for the 10 mg THC dose or five 5 mg capsules to be ingested for the 25 mg THC. Participants will be asked to complete PLR tests throughout the study day.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females 21 years of age or older
2. Females not of child-bearing potential, defined as those who have undergone a sterilization procedure (e.g. hysterectomy, bilateral oophorectomy, bilateral tubal ligation, complete endometrial ablation) or have been post-menopausal for at least 1 year prior to screening Or,

   Individuals of child-bearing potential must have a negative baseline urine pregnancy test and agree to use a medically approved method of birth control for the duration of the study. All hormonal birth control must have been in use for a minimum of three months. Acceptable methods of birth control include:
   1. Hormonal contraceptives including oral contraceptives, hormone birth control patch (Ortho Evra), vaginal contraceptive ring (NuvaRing), injectable contraceptives (Depo-Provera, Lunelle), or hormone implant (Norplant System)
   2. Double-barrier method
   3. Intrauterine devices
   4. Non-heterosexual lifestyle and agrees to use contraception if planning on changing to heterosexual partner(s)
   5. Vasectomy of partner at least 6 months prior to screening
   6. Abstinence and agrees to use contraception if planning on becoming sexually active during the study
3. Self-reported cannabis users based on the Cannabis Use Questionnaire who are familiar and experienced with THC's acute psychoactive effects from the doses and route of administration to be used in this study without previous severe adverse reactions after cannabis ingestion
4. Self-reported cannabis use at least 3x per month but no more than 3x per week
5. Agrees to abstain from cannabis use for 3 days prior to study visit
6. Willingness to complete all assessments associated with the study and agrees to safe transportation home
7. Provided voluntary, written, informed consent to participate in the study

Exclusion Criteria:

1. Individuals who are pregnant, breast feeding or planning to become pregnant during the study
2. Allergy, sensitivity, intolerance, or dietary restriction preventing consumption study products
3. Current and ongoing neurological or ophthalmological issue that could affect the retina (blindness, glaucoma, dry eyes, retinal diseases, pupil abnormalities, cataracts, sensitivity to bright lights)
4. History of surgery on eyes or retinas except for laser corneal surgery
5. Current or history of psychological disorders (e.g., schizophrenia and psychosis)
6. Current or history of any significant diseases of the gastrointestinal tract as assessed by the QI
7. Type I or Type II diabetes with diabetic retinopathy
8. Unstable metabolic disease or chronic diseases as assessed by the QI
9. Unstable hypertension. Treatment on a stable dose of medication for at least 3 months will be considered by the QI (see below)
10. Significant cardiovascular event in the past 6 months. Participants with no significant cardiovascular event on stable medication may be included after assessment by the QI on a case-by-case basis
11. History of or current diagnosis with kidney and/or liver diseases as assessed by the QI on a case-by-case basis, with the exception of history of kidney stones in participants who are symptom free for 6 months
12. Self-reported confirmation of current or pre-existing thyroid condition. Treatment on a stable dose of medication for at least 3 months will be considered by the QI
13. Major surgery in the past 3 months or individuals who have planned surgery during the course of the study. Participants with minor surgery will be considered on a case-by-case basis by the QI
14. Cancer, except skin basal cell carcinoma completely excised with no chemotherapy or radiation with a follow up that is negative. Volunteers with cancer in full remission for more than five years after diagnosis are acceptable
15. Individuals with an unstable autoimmune disease
16. Self-reported confirmation of a HIV-, Hepatitis B- and/or C-positive diagnosis as assessed by the QI
17. Alcohol or drug abuse within the last 12 months
18. Impairment from illicit drugs or alcohol during their study visit, as assessed by the QI or Sub-Investigator
19. Alcohol intake average of >2 standard drinks per day as assessed by the QI
20. Current use of prescribed and/or over-the-counter (OTC) medications, supplements, and/or consumption of food/drinks that may impact the efficacy and/or safety of the investigational product (see below)
21. Participation in other research studies 30 days prior to baseline, as assessed by the QI
22. Individuals who are cognitively impaired and/or who are unable to give informed consent
23. Any other condition or lifestyle factor, that, in the opinion of the QI, may adversely affect the participant's ability to complete the study or its measures or pose significant risk to the participant

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-05-22 (Actual); Primary Completion 2025-08 (Estimated); Study Completion 2025-08 (Estimated)

PRIMARY OUTCOMES:
The difference in change in Pupillary Light Reflex (PLR) measures between a smart phone-based test and NeuroLight pupillometer | T=0 to T=5 minutes
  The difference in change in PLR measures between a smart phone-based test and NeuroLight pupillometer in pupil size from time (T)=0 minutes (min) at T=5 min.
The difference in change in PLR measures between a smart phone-based test and NeuroLight pupillometer | T=0 to T=30 minutes
  The difference in change in PLR measures between a smart phone-based test and NeuroLight pupillometer in pupil size from time (T)=0 minutes (min) at T=30 min.
The difference in change in PLR measures between a smart phone-based test and NeuroLight pupillometer | T=0 to T=60 minutes
  The difference in change in PLR measures between a smart phone-based test and NeuroLight pupillometer in pupil size from time (T)=0 minutes (min) at T=60 min.
The difference in change in PLR measures between a smart phone-based test and NeuroLight pupillometer | T=0 to T=120 minutes
  The difference in change in PLR measures between a smart phone-based test and NeuroLight pupillometer in pupil size from time (T)=0 minutes (min) at T=120 min.
The difference in change in PLR measures between a smart phone-based test and NeuroLight pupillometer | T=0 to T=180 minutes
  The difference in change in PLR measures between a smart phone-based test and NeuroLight pupillometer in pupil size from time (T)=0 minutes (min) at T=180 min.
The difference in change in PLR measures between a smart phone-based test and NeuroLight pupillometer | T=0 to T=240 minutes
  The difference in change in PLR measures between a smart phone-based test and NeuroLight pupillometer in pupil size from time (T)=0 minutes (min) at T=240 min.
The difference in change in PLR measures between a smart phone-based test and NeuroLight pupillometer | T=0 to T=300 minutes
  The difference in change in PLR measures between a smart phone-based test and NeuroLight pupillometer in pupil size from time (T)=0 minutes (min) at T=300 min.
The difference in change in PLR measures between a smart phone-based test and NeuroLight pupillometer | T=0 to T=360 minutes
  The difference in change in PLR measures between a smart phone-based test and NeuroLight pupillometer in pupil size from time (T)=0 minutes (min) at T=360 min.
The difference in change in PLR measures between a smart phone-based test and NeuroLight pupillometer | T=0 to T=420 minutes
  The difference in change in PLR measures between a smart phone-based test and NeuroLight pupillometer in pupil size from time (T)=0 minutes (min) at T=420 min.
The difference in change in PLR measures between a smart phone-based test and NeuroLight pupillometer | T=0 to T=480 minutes
  The difference in change in PLR measures between a smart phone-based test and NeuroLight pupillometer in pupil size from time (T)=0 minutes (min) at T=480 min.
The difference in change in PLR measures between a smart phone-based test and NeuroLight pupillometer | T=0 to T=5 minutes
  The difference in change in pupil reflexes (absolute contraction and latency) between a smart phone-based test and NeuroLight pupillometer in pupil size from time (T)=0 minutes (min) at T=5 min.
The difference in change in PLR measures between a smart phone-based test and NeuroLight pupillometer | T=0 to T=30 minutes
  The difference in change in pupil reflexes (absolute contraction and latency) between a smart phone-based test and NeuroLight pupillometer from time (T)=0 minutes (min) at T=30 min.
The difference in change in PLR measures between a smart phone-based test and NeuroLight pupillometer | T=0 to T=60 minutes
  The difference in change in pupil reflexes (absolute contraction and latency) between a smart phone-based test and NeuroLight pupillometer from time (T)=0 minutes (min) at T=60 min.
The difference in change in PLR measures between a smart phone-based test and NeuroLight pupillometer | T=0 to T=120 minutes
  The difference in change in pupil reflexes (absolute contraction and latency) between a smart phone-based test and NeuroLight pupillometer from time (T)=0 minutes (min) at T=120 min.
The difference in change in PLR measures between a smart phone-based test and NeuroLight pupillometer | T=0 to T=180 minutes
  The difference in change in pupil reflexes (absolute contraction and latency) between a smart phone-based test and NeuroLight pupillometer from time (T)=0 minutes (min) at T=180 min.
The difference in change in PLR measures between a smart phone-based test and NeuroLight pupillometer | T=0 to T=240 minutes
  The difference in change in pupil reflexes (absolute contraction and latency) between a smart phone-based test and NeuroLight pupillometer from time (T)=0 minutes (min) at T=240 min.
The difference in change in PLR measures between a smart phone-based test and NeuroLight pupillometer | T=0 to T=300 minutes
  The difference in change in pupil reflexes (absolute contraction and latency) between a smart phone-based test and NeuroLight pupillometer from time (T)=0 minutes (min) at T=300 min.
The difference in change in PLR measures between a smart phone-based test and NeuroLight pupillometer | T=0 to T=360 minutes
  The difference in change in pupil reflexes (absolute contraction and latency) between a smart phone-based test and NeuroLight pupillometer from time (T)=0 minutes (min) at T=360 min.
The difference in change in PLR measures between a smart phone-based test and NeuroLight pupillometer | T=0 to T=480 minutes
  The difference in change in pupil reflexes (absolute contraction and latency) between a smart phone-based test and NeuroLight pupillometer from time (T)=0 minutes (min) at T=480 min.
The difference in change in PLR measures between a smart phone-based test and NeuroLight pupillometer | T=0 to T=5 minutes
  The difference in change in pupil activity as measured by pupillary unrest in ambient light (hippus) between a smart phone-based test and NeuroLight pupillometer in pupil size from time (T)=0 minutes (min) at T=5 min.
The difference in change in PLR measures between a smart phone-based test and NeuroLight pupillometer | T=0 to T=30 minutes
  The difference in change in pupil activity as measured by pupillary unrest in ambient light (hippus) between a smart phone-based test and NeuroLight pupillometer from time (T)=0 minutes (min) at T=30 min.
The difference in change in PLR measures between a smart phone-based test and NeuroLight pupillometer | T=0 to T=60 minutes
  The difference in change in pupil activity as measured by pupillary unrest in ambient light (hippus) between a smart phone-based test and NeuroLight pupillometer from time (T)=0 minutes (min) at T=60 min.
The difference in change in PLR measures between a smart phone-based test and NeuroLight pupillometer | T=0 to T=120 minutes
  The difference in change in pupil activity as measured by pupillary unrest in ambient light (hippus) between a smart phone-based test and NeuroLight pupillometer from time (T)=0 minutes (min) at T=120 min.
The difference in change in PLR measures between a smart phone-based test and NeuroLight pupillometer | T=0 to T=180 minutes
  The difference in change in pupil activity as measured by pupillary unrest in ambient light (hippus) between a smart phone-based test and NeuroLight pupillometer from time (T)=0 minutes (min) at T=180 min.
The difference in change in PLR measures between a smart phone-based test and NeuroLight pupillometer | T=0 to T=240 minutes
  The difference in change in pupil activity as measured by pupillary unrest in ambient light (hippus) between a smart phone-based test and NeuroLight pupillometer from time (T)=0 minutes (min) at T=240 min.
The difference in change in PLR measures between a smart phone-based test and NeuroLight pupillometer | T=0 to T=300 minutes
  The difference in change in pupil activity as measured by pupillary unrest in ambient light (hippus) between a smart phone-based test and NeuroLight pupillometer from time (T)=0 minutes (min) at T=300 min.
The difference in change in PLR measures between a smart phone-based test and NeuroLight pupillometer | T=0 to T=360 minutes
  The difference in change in pupil activity as measured by pupillary unrest in ambient light (hippus) between a smart phone-based test and NeuroLight pupillometer from time (T)=0 minutes (min) at T=360 min.
The difference in change in PLR measures between a smart phone-based test and NeuroLight pupillometer | T=0 to T=480 minutes
  The difference in change in pupil activity as measured by pupillary unrest in ambient light (hippus) between a smart phone-based test and NeuroLight pupillometer from time (T)=0 minutes (min) at T=480 min.

SECONDARY OUTCOMES:
The difference in change in reaction time | T= 0 at T=60 minutes
  The difference in change in reaction time as assessed by Dynavision from T= 0 at T=60 minutes
The difference in change in reaction time | T= 0 at T=120 minutes
  The difference in change in reaction time as assessed by Dynavision from T= 0 at T=120 min
The difference in change in reaction time | T= 0 at T=180 minutes
  The difference in change in reaction time as assessed by Dynavision from T= 0 at T=180 minutes
The difference in change in reaction time | T= 0 at T=240 minutes
  The difference in change in reaction time as assessed by Dynavision from T= 0 at T=240 minutes
The difference in change in reaction time | T= 0 at T=300 minutes
  The difference in change in reaction time as assessed by Dynavision from T= 0 at T=300 minutes
The difference in change in reaction time | T= 0 at T=360 minutes
  The difference in change in reaction time as assessed by Dynavision from T= 0 at T=360 min
The difference in change in reaction time | T= 0 at T=420 minutes
  The difference in change in reaction time as assessed by Dynavision from T= 0 at T=420 min
The difference in change in subjective drug effects | T=0 at T= 5 minutes
  The difference in change in subjective drug effects as assessed by the modified Drug Effects Questionnaire (DEQ) from T=0 at T= 5 min, on a scale of 1 to 10. Higher score indicates higher subjective drug effect.
The difference in change in subjective drug effects | T=0 at T=30 minutes
  The difference in change in subjective drug effects as assessed by the modified Drug Effects Questionnaire (DEQ) from T=0 at T=30 minutes, on a scale of 1 to 10. Higher score indicates higher subjective drug effect.
The difference in change in subjective drug effects | T=0 at T=60 minutes
  The difference in change in subjective drug effects as assessed by the modified Drug Effects Questionnaire (DEQ) from T=0 at T=60 minutes, on a scale of 1 to 10. Higher score indicates higher subjective drug effect.
The difference in change in subjective drug effects | T=0 at T=90 minutes
  The difference in change in subjective drug effects as assessed by the modified Drug Effects Questionnaire (DEQ) from T=0 at T=90 minutes, on a scale of 1 to 10. Higher score indicates higher subjective drug effect.
The difference in change in subjective drug effects | T=0 at T=120 minutes
  The difference in change in subjective drug effects as assessed by the modified Drug Effects Questionnaire (DEQ) from T=0 at T=120 minutes, on a scale of 1 to 10. Higher score indicates higher subjective drug effect.
The difference in change in subjective drug effects | T=0 at T=180 minutes
  The difference in change in subjective drug effects as assessed by the modified Drug Effects Questionnaire (DEQ) from T=0 at T=180 minutes, on a scale of 1 to 10. Higher score indicates higher subjective drug effect.
The difference in change in subjective drug effects | T=0 at T=240 minutes
  The difference in change in subjective drug effects as assessed by the modified Drug Effects Questionnaire (DEQ) from T=0 at T=240 minutes, on a scale of 1 to 10. Higher score indicates higher subjective drug effect.
The difference in change in subjective drug effects | T=0 at T=300 minutes
  The difference in change in subjective drug effects as assessed by the modified Drug Effects Questionnaire (DEQ) from T=0 at T=300 minutes, on a scale of 1 to 10. Higher score indicates higher subjective drug effect.
The difference in change in subjective drug effects | T=0 at T=360 minutes
  The difference in change in subjective drug effects as assessed by the modified Drug Effects Questionnaire (DEQ) from T=0 at T=360 minutes, on a scale of 1 to 10. Higher score indicates higher subjective drug effect.
The difference in change in subjective drug effects | T=0 at T=420 minutes
  The difference in change in subjective drug effects as assessed by the modified Drug Effects Questionnaire (DEQ) from T=0 at T=420 minutes, on a scale of 1 to 10. Higher score indicates higher subjective drug effect.
The difference in change in subjective drug effects | T=0 at T=480 minutes
  The difference in change in subjective drug effects as assessed by the modified Drug Effects Questionnaire (DEQ) from T=0 at T=480 minutes, on a scale of 1 to 10. Higher score indicates higher subjective drug effect.

OTHER OUTCOMES:
Clinically relevant post-emergent adverse events | T=0 to T=480 minutes
  Clinically relevant post-emergent adverse events at T=0 to T=480 minutes. Including via the modified Drug Effects Questionnaire (DEQ) from T=0 at T=480 minutes, on a scale of 1 to 10. Higher score indicates higher subjective drug effect.

CONTACTS AND LOCATIONS:
Overall Officials: David Crowley, MD, Principal Investigator — KGK Science Inc.
Locations (1):
- KGK Science Inc., London, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No